CLINICAL TRIAL: NCT06590324
Title: A Phase II, Multi-centre Open Label Study to Assess the Efficacy and Safety of Oral Apabetalone With Background Dapagliflozin in Subjects With Long -COVID-19 (Post-COVID-19 Conditions) and Type 2 Diabetes Mellitus (T2DM)
Brief Title: A Study of Apabetalone in Subjects With Long -COVID
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Resverlogix Corp (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RVX222-CS-025
Record Dates: First submitted 2024-08-26; First posted 2024-09-19 (Actual); Last update posted 2025-04-18 (Actual); Status verified 2025-04

CONDITIONS: Post-Acute COVID-19 Syndrome
MeSH Terms: conditions — Post-Acute COVID-19 Syndrome | interventions — apabetalone

STUDY DESIGN:
Intervention Model Description: Open Label Study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- apabetalone (Experimental): apabetalone selectively binds to the second bromodomain [BD2] of bromodomain extra terminal (BET) proteins, curbing the transcription of multiple disease associated genes that promote vascular inflammation, complement, acute phase response (APR), fibrosis, dyslipidemia, and vascular calcification.
  Interventions: Drug: Apabetalone

INTERVENTIONS:
Drug: Apabetalone — 100-mg capsule, twice daily oral administration with meals
  Other Names: RVX000222

SUMMARY:
This is an open label, multicentre, phase II clinical trial that aims to assess the efficacy and safety of oral Apabetalone with background dapagliflozin for up to 12 weeks in T2DM patients with a history of probable or confirmed SARS-CoV-2 infection, with symptoms within 3 months from the onset of COVID-19 that last for at least 2 months and cannot be explained by an alternative diagnosis.

DETAILED DESCRIPTION:
This is an open label, multicentre, phase II clinical trial that aims to assess the efficacy and safety of oral Apabetalone with background dapagliflozin for up to 12 weeks in T2DM patients with a history of probable or confirmed SARS-CoV-2 infection, with symptoms within 3 months from the onset of COVID-19 that last for at least 2 months and cannot be explained by an alternative diagnosis. Subjects will be receiving background therapy with dapagliflozin 10 mg daily.

In-person clinic visits will be used to collect data to assess the primary and secondary and exploratory endpoints. There will be 7 in-person visits.

After signing the informed consent form (ICF), and after all screening procedures have been performed, subject data will be reviewed by the Principal Investigator to determine subject eligibility. Eligible subjects will return for Visit 2 (Day 1) and assessments will be performed per the Schedule of Events. Subjects will be enrolled and treatment with Oral Apabetalone 100mg will be initiated. Subjects will be dispensed study drug to be administered at home with meals, twice daily.

ELIGIBILITY:
Inclusion Criteria:

1. Able and willing to provide written (signed and dated) informed consent before participation in the study, and to comply with scheduled visits, treatment plan, and other study-related procedures to complete the study.
2. Male or female subjects who are ≥ 18 years of age at Screening.
3. Documented diagnosis of T2DM (one or more of the following criteria must be met):

   1. Documented history of T2DM
   2. History of taking diabetes medication
   3. HbA1c ≥6.5% at Screening
4. Must be taking dapagliflozin as part of their diabetes medication, or, based on the Principal Investigator's judgment and indication, be willing to commence sponsor-provided dapagliflozin 10 mg daily for the duration of the study.
5. History of Long-COVID symptoms within 3 months from the onset of COVID-19 that have lasted for at least 2 months. Symptoms are listed in Long Covid Symptom Tool (LCST).
6. A Long Covid Impact Tool (LCIT) score of ≥ 30 at the Screening Visit and at Visit 2 (Day 1)
7. A negative SARS-CoV-2 test at the Screening Visit and at Visit 2 (Day 1)
8. Female subjects of childbearing potential and nonsterile male subjects with female partners of childbearing potential must agree to either remain abstinent or use highly effective non-hormonal methods of contraception throughout the study and at least 30 days after the last dose of study drug has been taken. Subjects must adhere to contraceptive use consistent with local regulations regarding the methods of contraception for those participating in clinical studies

   -

   Exclusion Criteria:
9. Subjects with chronic kidney disease (CKD) with an estimated glomerular filtration rate (eGFR) <25 mL/min/1.73 m2
10. New York Heart Association Class IV congestive heart failure
11. Evidence of cirrhosis from liver imaging or biopsy, a history of hepatic encephalopathy, esophageal or gastric varices, active hepatitis, or prior porta-caval shunt procedure; chronic liver diseases such as primary biliary cholangitis, untreated hemochromatosis, and primary sclerosing cholangitis
12. Subject meets any of the following laboratory criteria at Screening:

    * Alanine transaminase (ALT) or aspartate transaminase (AST) values > 1.5x the upper limit of normal (ULN)
    * Total bilirubin >1.5 × ULN.
    * Evidence of an active hepatitis B virus or hepatitis C virus infection
    * History of a positive test for human immunodeficiency virus (HIV)
13. Subjects taking concomitant cytochrome P450 3A4 strong inducers and/or strong inhibitors, or corticosteroid use >10 mg daily prednisone or equivalent.
14. Subjects who have received a COVID-19 vaccine or booster in the last 30 days prior to screening (Visit 1).
15. Subject who have participated in a clinical study and received any investigational medication within the last 30 days prior to screening (Visit 1).
16. Female subjects who are pregnant, planning to get pregnant, lactating/breastfeeding, or has a positive urine pregnancy test at the Screening Visit or prior to enrollment at the Day 1 visit.
17. Subjects whose safety may be compromised by study participation or are not, in the opinion of the investigator, able or willing to comply with the protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2025-04-15 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2026-03-30 (Estimated)

PRIMARY OUTCOMES:
patient acceptable symptom state (PASS) | 90 days
  The PASS assessment will consist of a single question phrased verbally by the delegated administrator as " Taking into account all your symptoms in daily life and your functional impairment, do you consider that your current state is satisfactory?". The response options are "Yes" or "No".

SECONDARY OUTCOMES:
Long COVID Symptom and Impact tools (LCST/LCIT) | 90 days
  These questionnaires will be presented to the subjects in paper format as a patient-reported instrument. Subjects indicate with a check mark which of the 53 symptoms they have experienced in the last 30 days. Symptoms are scored as the number checked by the subject (0-53) The disease's impact on their lives over the past 30 days is scored from the responses to 6 questions. Subjects will answer using a numeric scale ranging from 0 (no impact) to 10 (maximal impact)
Patient-Reported Outcomes Measurement Information System (PROMIS)-Fatigue Short Form 7a (SF-7a) | 90 days
  The PROMIS F-7a SF consists of seven items that measure both the experience of fatigue and the interference of fatigue on daily activities over the past week (NIH, 2007).
Baseline Dyspnea Index (BDI) & Transition Dyspnea Index (TDI) | 90 days
  The BDI and TDI are Interviewer-administered ratings of severity of dyspnea
Post-COVID-19 Functional Status (PCFS) Scale | 90 days
  The PCFS is an ordinal scale of 5 steps ranging from Grade 0 (No functional limitations) to Grade 4 (Severe functional limitations). This scale will be self-administered by the patient
DePaul Symptom Questionnaire - Post-Exertional Malaise Short Form (DSQ-PEM) | 90 days
  Post-exertional malaise (PEM) is a key symptom of chronic fatigue syndrome (CFS). Currently, five PEM-items from the DePaul Symptom Questionnaire (DSQ) will be used in this study to measure this symptom for patients with Post Covid Condition

OTHER OUTCOMES:
Biomarkers of inflammation | Days 1,14,30,60,90
  Change in biomarkers of inflammation from baseline. Assessed biomarkers will include Interferon (IFN): IFN-a, IFN-b, IFN-g, Interleukins (IL): IL-1a, IL-1b, IL-2, IL-4, IL-6, IL-7, IL-10, IL-10Rb, IL-12b, IL-13, IL-17, IL-18, IL-33, IP-10 and Tumor Necrosis Factor (TNF): TNF-a, TNF-b
biomarkers associated with Post-COVID-19 Condition and Chronic Fatigue Syndrome | Days 1,14,30,60,90
  Change in levels of Post-COVID-19 Condition and Chronic Fatigue Syndrome associated proteins. Assessed biomarkers will include:
  Immune system markers: CD4+, CD8+, CD27+, CD62L+, NKCD57+ and perforin+. Vascular biomarkers: Ang-2, D-dimer, Factor VIII:C, MMP-1, MMP-9, sICAM-1, sVCAM-1, VEGF, VWF:Ag, VWF:pp
blood transcriptome and plasma proteome and metabolomics | baseline in blood cell transcriptome at Day 1, Day 14 and change from baseline in plasma proteome at Days 1,14,30,60,90
  Change in RNA expression attributable to Post-COVID-19 Condition. Micro-RNA's assayed will include hsa-miR146a-5p, hsa-miR-126-3p and hsa-miR-223-3p. SARS-CoV-2-related host RNAs (ACE2/TMPRSS2 receptors, DPP4/FURIN proteases) and RNAs prototypical for memory B-cells and platelets will also be evaluated

CONTACTS AND LOCATIONS:
Overall Officials: Michael Sweeney, MD, Study Director — Resverlogix Corp
Locations (3):
- The Speciality Hospital, Amman, Jordan
- MNGHA- King Abdulaziz Hospital, Al Mubarraz, Saudi Arabia
- Al Kuwait Hospital, Dubai, Dubai, United Arab Emirates

IPD SHARING:
Plan to Share IPD: No